CLINICAL TRIAL: NCT02610712
Title: Clinical Trial of the Use of Ketamine in Treatment Resistant Depression
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Institute of Neurology and Neurosurgery, Mexico (Other)
Responsible Party: Principal Investigator, Rodrigo Pérez Esparza, Fourth-year Psychiatry Resident, National Institute of Neurology and Neurosurgery, Mexico
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 63/13
Record Dates: First submitted 2015-11-17; First posted 2015-11-20 (Estimated); Last update posted 2016-09-21 (Estimated); Status verified 2016-09

CONDITIONS: Depressive Disorder, Treatment-Resistant
Keywords: ketamine; treatment-resistant; depression; spectroscopy; neuroinflammation
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant; Depression; Neuroinflammatory Diseases | interventions — Ketamine

ARMS (1):
- TRD patients (Experimental): Treatment-Resistant (TRD) patients to receive intravenous ketamine at 0.5 mg/kg dose.
  Interventions: Drug: Ketamine

INTERVENTIONS:
Drug: Ketamine

SUMMARY:
The purpose of this study is to determine the efficacy of the use of intravenous low-dose ketamine in the treatment of treatment-resistant depression (TRD), as well as the changes in Glutamate neurotransmission and inflammatory serum markers.

DETAILED DESCRIPTION:
The purpose of this study is to determine the efficacy of the use of intravenous low-dose ketamine (0.5 mg/kg) in the treatment of treatment-resistant depression (TRD), as well as the changes in Glutamate neurotransmission measured by Magnetic Resonance Imaging Spectroscopy and inflammatory serum markers (IL-6, TNF-alpha).

ELIGIBILITY:
Inclusion Criteria:

* Treatment-Resistant Depression (Failure to respond to two or more trials of antidepressant monotherapy or failure to respond to four or more trials of different antidepressant therapies)
* Acceptance of participation via the informed consent

Exclusion Criteria:

* Psychiatric comorbidity (except anxiety related disorders)
* Substance abuse or dependence in the previous 3 months
* Evidence of structural abnormalities in brain imaging
* Pregnancy
* Previous hypersensitivity to ketamine
* Heart failure or insufficiency
* Familial or personal history of psychosis
* Glaucoma
* Major neurological disease
* Uncontrolled systemic arterial hypertension
* MRI contraindications
* Non-acceptance of participation via informed consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2014-05; Primary Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Hamilton Depression Rating Scale (HDRS) Score | Change from baseline HDRS Score at 24 hours

SECONDARY OUTCOMES:
Glutamate concentrations in the pregenual cingulate cortex (pgACC) | Change from baseline Glutamate concentrations in the pgACC at 24 hours
  Glutamate concentrations in the pregenual cingulate cortex measured by Magnetic Resonance Spectroscopy
Interleukin-1 (IL-1) and Tumoral Necrosis Factor-alpha (TNF-alpha) serum concentrations | Change from baseline IL-1 and TNF-alpha serum concentrations from baseline at 24 hours
  Interleukin-1 and Tumoral Necrosis Factor-alpha concentrations in serum measured by ELISA

CONTACTS AND LOCATIONS:
Overall Officials: Rodrigo Pérez-Esparza, MD, Principal Investigator — National Institute of Neurology and Neurosurgery, Mexico; Jesús Ramírez-Bermúdez, MD, MSc, Principal Investigator — National Institute of Neurology and Neurosurgery, Mexico
Locations (1):
- National Institute of Neurology and Neurosurgery, Mexico City, Mexico City, Mexico

REFERENCES:
- [Background] Berman RM, Cappiello A, Anand A, Oren DA, Heninger GR, Charney DS, Krystal JH. Antidepressant effects of ketamine in depressed patients. Biol Psychiatry. 2000 Feb 15;47(4):351-4. doi: 10.1016/s0006-3223(99)00230-9. PMID 10686270
- [Background] DiazGranados N, Ibrahim LA, Brutsche NE, Ameli R, Henter ID, Luckenbaugh DA, Machado-Vieira R, Zarate CA Jr. Rapid resolution of suicidal ideation after a single infusion of an N-methyl-D-aspartate antagonist in patients with treatment-resistant major depressive disorder. J Clin Psychiatry. 2010 Dec;71(12):1605-11. doi: 10.4088/JCP.09m05327blu. Epub 2010 Jul 13. PMID 20673547
- [Background] Valentine GW, Mason GF, Gomez R, Fasula M, Watzl J, Pittman B, Krystal JH, Sanacora G. The antidepressant effect of ketamine is not associated with changes in occipital amino acid neurotransmitter content as measured by [(1)H]-MRS. Psychiatry Res. 2011 Feb 28;191(2):122-7. doi: 10.1016/j.pscychresns.2010.10.009. Epub 2011 Jan 12. PMID 21232924
- [Background] Zarate CA Jr, Brutsche NE, Ibrahim L, Franco-Chaves J, Diazgranados N, Cravchik A, Selter J, Marquardt CA, Liberty V, Luckenbaugh DA. Replication of ketamine's antidepressant efficacy in bipolar depression: a randomized controlled add-on trial. Biol Psychiatry. 2012 Jun 1;71(11):939-46. doi: 10.1016/j.biopsych.2011.12.010. Epub 2012 Jan 31. PMID 22297150
- [Background] Zarate CA Jr, Singh JB, Carlson PJ, Brutsche NE, Ameli R, Luckenbaugh DA, Charney DS, Manji HK. A randomized trial of an N-methyl-D-aspartate antagonist in treatment-resistant major depression. Arch Gen Psychiatry. 2006 Aug;63(8):856-64. doi: 10.1001/archpsyc.63.8.856. PMID 16894061
- [Background] Diazgranados N, Ibrahim L, Brutsche NE, Newberg A, Kronstein P, Khalife S, Kammerer WA, Quezado Z, Luckenbaugh DA, Salvadore G, Machado-Vieira R, Manji HK, Zarate CA Jr. A randomized add-on trial of an N-methyl-D-aspartate antagonist in treatment-resistant bipolar depression. Arch Gen Psychiatry. 2010 Aug;67(8):793-802. doi: 10.1001/archgenpsychiatry.2010.90. PMID 20679587
- [Background] Horn DI, Yu C, Steiner J, Buchmann J, Kaufmann J, Osoba A, Eckert U, Zierhut KC, Schiltz K, He H, Biswal B, Bogerts B, Walter M. Glutamatergic and resting-state functional connectivity correlates of severity in major depression - the role of pregenual anterior cingulate cortex and anterior insula. Front Syst Neurosci. 2010 Jul 15;4:33. doi: 10.3389/fnsys.2010.00033. eCollection 2010. PMID 20700385
- [Background] Murrough JW, Iosifescu DV, Chang LC, Al Jurdi RK, Green CE, Perez AM, Iqbal S, Pillemer S, Foulkes A, Shah A, Charney DS, Mathew SJ. Antidepressant efficacy of ketamine in treatment-resistant major depression: a two-site randomized controlled trial. Am J Psychiatry. 2013 Oct;170(10):1134-42. doi: 10.1176/appi.ajp.2013.13030392. PMID 23982301
- [Background] Musazzi L, Treccani G, Mallei A, Popoli M. The action of antidepressants on the glutamate system: regulation of glutamate release and glutamate receptors. Biol Psychiatry. 2013 Jun 15;73(12):1180-8. doi: 10.1016/j.biopsych.2012.11.009. Epub 2012 Dec 28. PMID 23273725
- [Background] Luykx JJ, Laban KG, van den Heuvel MP, Boks MP, Mandl RC, Kahn RS, Bakker SC. Region and state specific glutamate downregulation in major depressive disorder: a meta-analysis of (1)H-MRS findings. Neurosci Biobehav Rev. 2012 Jan;36(1):198-205. doi: 10.1016/j.neubiorev.2011.05.014. Epub 2011 Jun 6. PMID 21672551
- [Background] Stone JM, Dietrich C, Edden R, Mehta MA, De Simoni S, Reed LJ, Krystal JH, Nutt D, Barker GJ. Ketamine effects on brain GABA and glutamate levels with 1H-MRS: relationship to ketamine-induced psychopathology. Mol Psychiatry. 2012 Jul;17(7):664-5. doi: 10.1038/mp.2011.171. Epub 2012 Jan 3. No abstract available. PMID 22212598
- [Background] Miller AH, Maletic V, Raison CL. Inflammation and its discontents: the role of cytokines in the pathophysiology of major depression. Biol Psychiatry. 2009 May 1;65(9):732-41. doi: 10.1016/j.biopsych.2008.11.029. Epub 2009 Jan 15. PMID 19150053
- [Background] Dowlati Y, Herrmann N, Swardfager W, Liu H, Sham L, Reim EK, Lanctot KL. A meta-analysis of cytokines in major depression. Biol Psychiatry. 2010 Mar 1;67(5):446-57. doi: 10.1016/j.biopsych.2009.09.033. Epub 2009 Dec 16. PMID 20015486